CLINICAL TRIAL: NCT00118248
Title: A Phase II Trial of 17-Allylaminogeldanamycin (17AAG) in Advanced Medullary and Differentiated Thyroid Carcinoma
Brief Title: Tanespimycin in Treating Patients With Inoperable Locoregionally Advanced or Metastatic Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00063; NCI-2009-00063 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); JHOC-B/06/174; NCI-6482; JHOC-JS0652; CDR0000433150; MC0476 (Other: Mayo Clinic); 6482 (Other: CTEP); N01CM62205 (NIH); P30CA015083 (NIH); N01CM62207 (NIH); NCT01646944 (obsolete NCT alias); NCT01664351 (obsolete NCT alias)
Record Dates: First submitted 2005-07-08; First posted 2005-07-11 (Estimated); Results first posted 2014-05-06 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2016-12

CONDITIONS: Recurrent Thyroid Cancer; Stage IV Follicular Thyroid Cancer; Stage IV Papillary Thyroid Cancer; Thyroid Gland Medullary Carcinoma
MeSH Terms: conditions — Thyroid Neoplasms; Adenocarcinoma, Follicular; Thyroid Cancer, Papillary; Carcinoma, Medullary | interventions — tanespimycin

ARMS (1):
- Treatment (chemotherapy) (Experimental): Patients receive tanespimycin IV over 2-6 hours on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: tanespimycin

INTERVENTIONS:
Drug: tanespimycin — Given IV
  Other Names: 17-AAG

SUMMARY:
This phase II trial is studying how well tanespimycin works in treating patients with inoperable locoregionally advanced or metastatic thyroid cancer. Drugs used in chemotherapy, such as tanespimycin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the 1-year treatment failure rate in patients with inoperable locoregionally advanced or metastatic medullary or differentiated thyroid carcinoma treated with 17-N-allylamino-17-demethoxygeldanamycin (17-AAG) (tanespimycin).

SECONDARY OBJECTIVES:

I. Determine the toxicity of this drug in these patients. Determine the 1-year progression-free rate in patients treated with this drug.

II. Determine the response rate and duration of response in patients treated with this drug.

III. Determine the time to treatment failure and time to subsequent therapy in patients treated with this drug.

IV. Determine the time to disease progression and overall survival of patients treated with this drug.

V. Correlate the incidence rate of RAS, RAF, and RET mutations with clinical outcome in patients treated with this drug.

OUTLINE: This is a multicenter study. Patients are stratified according to type of thyroid carcinoma (medullary vs differentiated).

Patients receive tanespimycin intravenously (IV) over 2-6 hours on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months until disease progression and then every 6 months for up to 3 years from study entry.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of thyroid carcinoma of 1 of the following types:

  * Medullary
  * Differentiated

    * Iodine I 131-resistant disease, defined as failure to incorporate and/or progression of measurable disease after treatment with iodine I 131
* Inoperable locoregionally advanced or metastatic disease
* Measurable disease, defined as ≥ 1 lesion ≥ 2.0 cm by conventional techniques OR ≥ 1.0 cm by spiral CT scan
* No active CNS metastases
* Performance status - ECOG 0-2
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL
* Bilirubin ≤ normal
* Alkaline phosphatase ≤ 2.5 times upper limit of normal (ULN)
* AST ≤ 1.5 times ULN
* Creatinine ≤ 1.5 times ULN
* QTc < 450 msec for male patients (470 msec for female patients)
* LVEF > 40% by MUGA
* DLCO ≥ 80%
* No cardiac symptoms ≥ grade 2
* No active ischemic heart disease within the past year
* No congenital long QT syndrome
* No left bundle branch block
* No history of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation ≥ 3 beats in a row)
* No myocardial infarction within the past year
* No New York Heart Association class III or IV congestive heart failure
* No poorly controlled angina
* No history of angina (of any sort) within the past 6 months
* No history of uncontrolled dysrhythmias or requiring antiarrhythmic drugs
* No history of cardiac toxicity after treatment with anthracyclines (e.g., doxorubicin hydrochloride, daunorubicin hydrochloride, mitoxantrone hydrochloride, bleomycin, or carmustine)
* No other significant cardiac disease
* No uncontrolled infection
* No history of serious allergic reaction to eggs
* No pulmonary symptoms ≥ grade 2
* No symptomatic pulmonary disease requiring medication including the following:

  * Dyspnea on or off exertion
  * Paroxysmal nocturnal dyspnea
  * Oxygen requirement
  * Significant pulmonary disease (e.g., chronic obstructive/restrictive pulmonary disease)
* No home oxygen need meeting the Medicare criteria
* No history of pulmonary toxicity after treatment with anthracyclines (e.g., doxorubicin hydrochloride, daunorubicin hydrochloride, mitoxantrone hydrochloride, bleomycin, or carmustine)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or noninvasive carcinoma
* No active seizure disorder
* More than 4 weeks since prior and no concurrent immunotherapy
* More than 4 weeks since prior biologic therapy
* No concurrent routine or prophylactic colony-stimulating factors (e.g., filgrastim [G-CSF] or sargramostim [GM-CSF])
* More than 4 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosoureas) and recovered
* No other concurrent chemotherapy
* See Disease Characteristics
* More than 4 weeks since prior and no concurrent radiotherapy
* More than 4 weeks since prior radiopharmaceuticals
* No prior radiotherapy to > 25% of bone marrow
* No prior radiotherapy that potentially included the heart in the field (i.e., mantle) or chest
* More than 4 weeks since prior therapeutic surgery for the tumor
* More than 3 months since prior sublingual nitroglycerin
* No other concurrent investigational ancillary therapy
* Concurrent CYP3A4 inhibitors allowed
* No concurrent medications that prolong or may prolong QTc interval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2004-12; Primary Completion 2009-08 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Moley, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From February 2005 thru April 2009, 41 participants were accrued to the this study.
  The study was closed to enrollment in July, 2009 due to a slow accrual rate.
Pre-assignment Details: From February 2005 thru February 2009, 17 participants were accrued to the Advanced Medullary Thyroid Carcinoma group. From February 2008 thru April 2009, 24 participants were accrued to the Differentiated Thyroid Carcinoma group.
Groups:
- Advanced Medullary Thyroid Carcinoma Group; Differentiated Thyroid Carcinoma: Patients receive 220 mg/m^2 tanespimycin IV over 2-6 hours on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Advanced Medullary Thyroid Carcinoma Group | Differentiated Thyroid Carcinoma
Started | 17 | 24
Completed | 17 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Advanced Medullary Thyroid Carcinoma Group | Differentiated Thyroid Carcinoma | Total
Number analyzed (Participants) | 17 | 24 | 41
Age, Continuous [Median (Full Range); unit: years] | 56 [33 to 70] | 61 [34 to 80] | 60 [33 to 80]
Gender [Count of Participants; unit: Participants]
  Female | 5 | 11 | 16
  Male | 12 | 13 | 25
Region of Enrollment [Number; unit: participants]
  United States | 17 | 24 | 41

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Have Remained on Treatment and Progression-free at Least One Year After Start of 17-AAG (Tanespimycin)
Description: The one-year treatment failure free rate is 100% times the proportion of eligible patients who remain on treatment and are progression-free at least one year after treatment start. A 90% confidence interval for the one year treatment failure free rate was constructed using the properties of the binomial confidence interval.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Patients that are not classified as having a progression are termed progression-free.
Time Frame: 1 year
Population: All patients were evaluable for this endpoint in this group.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Advanced Medullary Thyroid Carcinoma Group | Differentiated Thyroid Carcinoma
Number analyzed (Participants) | 17 | 24
percentage of participants | 5.9 [0.3 to 25.0] | 12.5 [3.5 to 29.2]

2. Secondary Outcome: Overall Response
Description: The number of responses were categorized and summarized independently within each of the patient groups. Participants were evaluated using Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.0.
  Complete Response (CR): Disappearance of all lesions.
  Partial Response (PR): At least a 30% decrease in the sum of the longest dimension (LD) of target lesions taking as reference the baseline sum LD.
Time Frame: Baseline, every 3 courses, and at the end of treatment study
Population: All participants were evaluated for response.
Measure: Number; unit: participants
Arm/Group | Advanced Medullary Thyroid Carcinoma Group | Differentiated Thyroid Carcinoma
Number analyzed (Participants) | 17 | 24
participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 1 | 0

3. Secondary Outcome: Progression-Free Survival
Description: Defined as the time from registration to the date of progression or death due to any cause. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Patients that are not classified as having a progression are termed progression-free. Estimated using the Kaplan-Meier method.
Time Frame: Every 3 months for up to 3 years
Population: All participants were evaluable for this endpoint.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Advanced Medullary Thyroid Carcinoma Group | Differentiated Thyroid Carcinoma
Number analyzed (Participants) | 17 | 24
months | 6.4 [2.7 to 17.2] | 4.1 [2.2 to 8.7]

4. Secondary Outcome: Overall Survival
Description: Defined as the time from registration to date of last follow-up or death due to any cause. Estimated using the Kaplan-Meier method.
Time Frame: Every 3 months until progression, and then every 6 months up to 3 years
Population: All patients were evaluable for this endpoint.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Advanced Medullary Thyroid Carcinoma Group | Differentiated Thyroid Carcinoma
Number analyzed (Participants) | 17 | 24
years | 2.1 [0.67 to 3.1] | 1.5 [0.73 to 3.5]

5. Secondary Outcome: Toxicity
Description: Defined as the number of participants reporting grade 3 or higher adverse events that are classified as either possibly, probably, or definitely related to study treatment. Determined using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
Time Frame: Every 3 courses during treatment (median cycle number was 5 with a maximum of 38 cycles)
Population: All participants were evaluable for this endpoint.
Measure: Number; unit: participants
Arm/Group | Advanced Medullary Thyroid Carcinoma Group | Differentiated Thyroid Carcinoma
Number analyzed (Participants) | 17 | 24
participants
  Grade 3 or Higher | 4 | 9
  Grade 4 or Higher | 3 | 0
  Grade 5 | 1 | 0

ADVERSE EVENTS:
Groups:
- All Patients: Patients receive 220 mg/m^2 tanespimycin IV over 2-6 hours on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 13/41
Other Adverse Events (participants affected / at risk) | 39/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=41)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Edema limbs (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (3)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=41)
Hemoglobin decreased (Blood and lymphatic system disorders) | 24 (104)
Lymph node pain (Blood and lymphatic system disorders) | 2 (3)
Cardiac disorder (Cardiac disorders) | 1 (1)
Ear disorder (Ear and labyrinth disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (11)
Tinnitus (Ear and labyrinth disorders) | 1 (12)
Hypothyroidism (Endocrine disorders) | 1 (4)
Photophobia (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (13)
Diarrhea (Gastrointestinal disorders) | 25 (63)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (6)
Dysphagia (Gastrointestinal disorders) | 6 (17)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 22 (93)
Tooth disorder (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 11 (23)
Chest pain (General disorders) | 1 (1)
Chills (General disorders) | 4 (6)
Edema limbs (General disorders) | 4 (15)
Fatigue (General disorders) | 26 (72)
Fever (General disorders) | 3 (4)
Localized edema (General disorders) | 1 (1)
Pain (General disorders) | 3 (4)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (5)
Bruising (Injury, poisoning and procedural complications) | 2 (6)
Alanine aminotransferase increased (Investigations) | 21 (74)
Alkaline phosphatase increased (Investigations) | 19 (71)
Aspartate aminotransferase increased (Investigations) | 18 (64)
Blood bilirubin increased (Investigations) | 9 (41)
Creatinine increased (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 6 (17)
Leukocyte count decreased (Investigations) | 9 (42)
Lymphocyte count decreased (Investigations) | 10 (26)
Neutrophil count decreased (Investigations) | 5 (11)
Platelet count decreased (Investigations) | 3 (5)
Weight loss (Investigations) | 4 (5)
Anorexia (Metabolism and nutrition disorders) | 7 (12)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 6 (9)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Serum albumin decreased (Metabolism and nutrition disorders) | 2 (2)
Serum calcium decreased (Metabolism and nutrition disorders) | 4 (6)
Serum calcium increased (Metabolism and nutrition disorders) | 4 (4)
Serum glucose decreased (Metabolism and nutrition disorders) | 2 (3)
Serum potassium decreased (Metabolism and nutrition disorders) | 5 (7)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 2 (3)
Serum sodium increased (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (7)
Arthritis (Musculoskeletal and connective tissue disorders) | 5 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (9)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (9)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (17)
Neck pain (Musculoskeletal and connective tissue disorders) | 5 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 4 (22)
Dysgeusia (Nervous system disorders) | 5 (8)
Headache (Nervous system disorders) | 6 (11)
Peripheral motor neuropathy (Nervous system disorders) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (15)
Anxiety (Psychiatric disorders) | 6 (18)
Depression (Psychiatric disorders) | 6 (17)
Insomnia (Psychiatric disorders) | 6 (19)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (30)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15 (41)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (6)
Body odor (Skin and subcutaneous tissue disorders) | 7 (15)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 2 (3)
Sweating (Skin and subcutaneous tissue disorders) | 4 (10)
Flushing (Vascular disorders) | 2 (3)
Hot flashes (Vascular disorders) | 1 (3)
Hypertension (Vascular disorders) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less